CLINICAL TRIAL: NCT06497322
Title: Effectiveness of High-intensity Interval Training During Neoadjuvant Immunochemotherapy on Complete Remission in Patients With Triple-negative Breast Cancer
Brief Title: Exercise Intervention in Women Diagnosed With Triple-negative Breast Cancer Receiving Oncologic Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Cologne (Other)
Collaborators: St. Elisabeth Krankenhaus Köln-Hohenlind (Unknown)
Responsible Party: Principal Investigator, Freerk Bauman, Prof.dr. Freerk T. Baumann, University Hospital of Cologne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No. 13-050
Record Dates: First submitted 2024-06-25; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
Keywords: Exercise; Immunotherapy; Oxygen uptake; CT scan; Blood markers
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled intervention (1:1 randomization). Specifically, 1 control group (usual care) and 1 intervention group (HIIT aerobic training), both receiving neoadjuvant therapy (immunochemotherapy) by infusion, as follows; Paclitaxel 80mg/m2 q1w x12, carboplatin 1.5 AUC q1w x12, pembrolizumab 200mg q3w x4, followed by epirubicin 90mg/ m2 q3w x 4, cyclophosphamide 600mg m2 q3w x 4, pembrolizumab 200mg q3w x 4. The intervention period (oncologic therapy + exercise intervention) is approximately 6 months (including screening phase and baseline data collection, tao), data collection after three months (ta1), after completion of neoadjuvant therapy (~six months ta2), during which participants will complete the exercise intervention + oncologic treatment on site. Surgery will take place 2-3 weeks later.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): All women in the experimental group receive standardized high-intensity interval training over a period of 6 months in combination with neoadjuvant therapy (immunochemotherapy). The individual training sessions are guided and monitored by qualified exercise therapists, taking into account the side effects of ongoing treatment. Each training session will last about one hour, with the effective training time being 30 minutes. Bike training begins 1 hour before neoadjuvant therapy and then at the same time of day between therapies. The TNBC patients start with 5 minutes of cycling followed by 3 × 3 - minute HIIT training sequences, constantly alternating: i) 30 s at 90% of maximal PO (70 rpm for 30 s) and ii) 30 s of light pedaling at 20% of PO). The training session will be concluded with a 5-min cool-down cycling (easy pedaling) and stretching. This protocol will be performed twice a week throughout the study.
  Interventions: Other: Exercise intervention - High intensity interval training on a cycle-ergometer
- Control group (No Intervention): The control group will receive the standard care during their neoadjuvant therapy (immunochemotherapy) over a 6-month period.

INTERVENTIONS:
Other: Exercise intervention - High intensity interval training on a cycle-ergometer — The experimental group starts with 5 minutes of unloaded cycling, followed by 3 × 3-minute HIIT training sequences alternating between: i) 30 seconds at 90% of maximal PO (70 rpm for 30 seconds) and ii) 30 seconds of light pedaling at 20% of PO). Recent work suggests that this high-intensity approach to aerobic exercise is feasible and safe, even during acute oncology treatment. The HIIT sequences are interspersed with two 3-minute cycling sessions at moderate intensity. The training session will be concluded with a 5-minute cool-down by cycling (light pedaling) and stretching. This protocol will be performed twice a week throughout the study, and all patients who reach an 80% adherence threshold for the exercise intervention will be included in the final analysis.
  Arms: Experimental group

SUMMARY:
In this randomized, controlled, prospective, two-arm intervention study, the investigators plan to investigate the effects of high-intensity interval training in women diagnosed with triple-negative breast cancer. Breast cancer is one of the most common cancers and one of the leading causes of cancer-related deaths worldwide. Among the different subtypes, triple-negative breast cancer accounts for about 15-20% of all breast cancer cases and is characterized by a more aggressive clinical course. Recent results indicate that the percentage of patients with a pathologic complete response was 13% higher in the chemotherapy-immunotherapy group (by 64.8%) than in the placebo-chemotherapy group (51.2). High-intensity interval training has a positive effect on the immune system, suggesting that it may improve the efficacy of chemo-immunotherapy, leading to a higher rate of pathologic complete response (pCR) in patients with newly diagnosed triple-negative breast cancer. In addition to the immunomodulatory effects, this exercise model could boost microvascular perfusion, thereby improving tumor perfusion, enhancing chemo-immunotherapy and leading to better outcomes.

DETAILED DESCRIPTION:
Recent clinical trials showed promising results in patients with triple negative breast cancer (TNBC) who received four cycles of pembrolizumab (at a dose of 200 mg) every three weeks + standard chemotherapy, compared to patients who received placebo + chemotherapy alone. Importantly, the overall risk of disease progression that precluded surgery, local or distant recurrence, occurrence of a second primary cancer, or death from any cause was 37% lower with pembrolizumab chemotherapy compared to placebo chemotherapy. Exercise training is a supportive multi-effect strategy with the ability to influence multiple organ systems. There is growing epidemiologic evidence that a physically active lifestyle is associated with a lower risk of developing cancer, particularly colon and breast cancer. Recent preclinical studies suggest that exercise can control and attenuate the growth of tumor cells. Therefore, exercise could be a potential means to increase the rate of pCR in cancer patients in general. High-intensity interval training resulted in higher cardiorespiratory fitness levels, particularly in breast cancer and lung patients who exercised for at least 8 weeks, with a significant improvement (from 2.40 to 4.19 mL-min-1-kg-1) observed compared to control groups. The aim of this study is to investigate the effects of HIIT training on immune system response and pCR rates (most commonly defined as complete eradication of the tumor as a surrogate parameter for good prognosis) during neoadjuvant immunochemotherapy in women with TNBC. The working hypothesis is that HIIT training would activate the immune system and enhance the combination of neoadjuvant treatment, leading to higher rates of pCR in the aerobic group compared to the usual treatment group. Thus, this exercise model may also promote microvascular perfusion, improve tumor perfusion, and potentially lead to more favorable outcomes in neoadjuvant therapy, increasing the efficacy of systemic treatments and allowing for better therapeutic outcomes. The researchers support the idea that high-intensity aerobic exercise may at least partially challenge the large heterogeneity in response to medical treatment in women with a first diagnosis of TNBC and lead to higher response rates in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of histologically verified triple-negative breast cancer (TNBC) measurable by ultrasound imaging
* Stage of disease: T1c and nodal status N1-2 or Stage T2-4 and nodal status N0-2
* Deemed eligible for intended treatment with Paclitaxel 80mg/m2 q1w x12, Carboplatin 1,5 AUC q1w x12, Pembrolizumab 200mg q3w x4 followed by Epirubicin 90mg/ m2 q3w x 4, Cyclophosphamid 600mg m2 q3w x 4, Pembrolizumab 200mg q3w x 4; by the treating physician
* Treatment in curative intent with life expectancy ≥ 3 months
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 12 months after the last dose of study treatment for participants who have received cyclophosphamide, and 6 months after the last dose of study treatment for participants who did not.
* Sufficient German language skills;

Exclusion Criteria:

* History of invasive malignancy ≤2 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Any history of previous systemic treatment for TNBC;
* Any diseases that do not allow sports activity, such as:

  * Clinically-manifest heart failure (NYHA III-IV);
  * Respiratory partial or global insufficiency;
  * Permanent thrombocytopenia <10,000/µl, e.g., refractory autoimmune thrombocytopenia;
  * Congenital or acquired thrombocytopathies or coagulation disorders.
  * Symptomatic CHD (clearance certificate required, stress ECG and cardiac ultrasound recommended if necessary);
* Participation in another exercise study;

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission of the tumor (pCR); | After completion of neoadjuvant therapy and after surgery (6 months from study onset)
  The absence of residual invasive cancer of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy (i.e., ypT0/Tis ypN0 in the current AJCC staging system)

SECONDARY OUTCOMES:
Mamma- Ultrasound (the overall response rate of tumor mass); | Baseline (prior to any data collection or therapy administration), and every three weeks during neoadjuvant chemotherapy
  Ultrasound imaging
Progression free survival and Overall survival | Epidemiological data collected during the study and three years afterwards
  Clinically relevant data
Cardiorespiratory fitness | At baseline (prior to any data collection or therapy administration), three months after baseline, and six months after baseline (following completion of neoadjuvant therapy)
  Measures of oxygen uptake via CPET
OCTA - optical coherence tomography angiography | At baseline (prior to any data collection or therapy administration) and after the completion of neoadjuvant therapy (most commonly 6 months)
  Measure of blood vessel compliance for the eye
Biomarkers of immune response | At baseline (prior to any data collection or therapy administration) and after the completion of neoadjuvant therapy (most commonly 6 months)
  Blood sampling to measure i) Longitudinal dynamics of soluble biomarkers such as e.g. CRP (mg/dL); ii) Longitudinal dynamics of blood counts such as e.g. leukocytes (cells/uL); iii) Longitudinal dynamics of immune cell subsets measured by flow-cytometry such as e.g. activated T-cells (CD8+HLA-DR+)
Quality of life, cancer-related fatigue, treatment tolerance and side-effects; physical activity behavior. | Baseline, and after the completion of neoadjuvant therapy (most likely 6 months after baseline)
  Questionnaire items (0 - 100 scale, with 0 being lower and 100 being the higher, positive outcome);

CONTACTS AND LOCATIONS:
Overall Officials: Freerk T Baumann, PhD, Principal Investigator — University Hospital of Cologne
Locations (1):
- University Hospital of Cologne and St. Elizabeth Hospital, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
All patient-related data is collected in pseudonymized form. The procedure for pseudonymization will be as follows: The investigator will receive a patient identification form in his study folder. All study patients must be entered there with their full name, date of birth, study initials, and patient documentation sheet number. The patient identification list will be kept separate from the documentation records at the center. This list must be kept completely confidential and must not leave the study center. The patient identification list must be archived for 10 years after the end of the study and then destroyed. Data processing and data management is carried out by the University Hospital Cologne. It stores all changes to the data in an audit trail and has a study-specific customizable user and role concept. The database is integrated into a general IT infrastructure and security concept with firewall and backup system.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After data collection and analysis are completed.
Access Criteria: Upon reasonable request to the study principal investigator.

REFERENCES:
- [Result] Schmid P, Cortes J, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Foukakis T, Fasching PA, Cardoso F, Untch M, Jia L, Karantza V, Zhao J, Aktan G, Dent R, O'Shaughnessy J; KEYNOTE-522 Investigators. Pembrolizumab for Early Triple-Negative Breast Cancer. N Engl J Med. 2020 Feb 27;382(9):810-821. doi: 10.1056/NEJMoa1910549. PMID 32101663
- [Result] Cortes J, Rugo HS, Cescon DW, Im SA, Yusof MM, Gallardo C, Lipatov O, Barrios CH, Perez-Garcia J, Iwata H, Masuda N, Torregroza Otero M, Gokmen E, Loi S, Guo Z, Zhou X, Karantza V, Pan W, Schmid P; KEYNOTE-355 Investigators. Pembrolizumab plus Chemotherapy in Advanced Triple-Negative Breast Cancer. N Engl J Med. 2022 Jul 21;387(3):217-226. doi: 10.1056/NEJMoa2202809. PMID 35857659
- [Result] Sheinboim D, Parikh S, Manich P, Markus I, Dahan S, Parikh R, Stubbs E, Cohen G, Zemser-Werner V, Bell RE, Ruiz SA, Percik R, Brenner R, Leibou S, Vaknine H, Arad G, Gerber Y, Keinan-Boker L, Shimony T, Bikovski L, Goldstein N, Constantini K, Labes S, Mordechai S, Doron H, Lonescu A, Ziv T, Nizri E, Choshen G, Eldar-Finkelman H, Tabach Y, Helman A, Ben-Eliyahu S, Erez N, Perlson E, Geiger T, Ben-Zvi D, Khaled M, Gepner Y, Levy C. An Exercise-Induced Metabolic Shield in Distant Organs Blocks Cancer Progression and Metastatic Dissemination. Cancer Res. 2022 Nov 15;82(22):4164-4178. doi: 10.1158/0008-5472.CAN-22-0237. PMID 36084256
- [Result] Wolin KY, Yan Y, Colditz GA. Physical activity and risk of colon adenoma: a meta-analysis. Br J Cancer. 2011 Mar 1;104(5):882-5. doi: 10.1038/sj.bjc.6606045. Epub 2011 Feb 8. PMID 21304525
- [Result] Wu Y, Zhang D, Kang S. Physical activity and risk of breast cancer: a meta-analysis of prospective studies. Breast Cancer Res Treat. 2013 Feb;137(3):869-82. doi: 10.1007/s10549-012-2396-7. Epub 2012 Dec 30. PMID 23274845
- [Result] Sanft T, Harrigan M, McGowan C, Cartmel B, Zupa M, Li FY, Ferrucci LM, Puklin L, Cao A, Nguyen TH, Neuhouser ML, Hershman DL, Basen-Engquist K, Jones BA, Knobf T, Chagpar AB, Silber A, Tanasijevic A, Ligibel JA, Irwin ML. Randomized Trial of Exercise and Nutrition on Chemotherapy Completion and Pathologic Complete Response in Women With Breast Cancer: The Lifestyle, Exercise, and Nutrition Early After Diagnosis Study. J Clin Oncol. 2023 Dec 1;41(34):5285-5295. doi: 10.1200/JCO.23.00871. Epub 2023 Sep 1. PMID 37656930
- [Result] Lavin-Perez AM, Collado-Mateo D, Mayo X, Humphreys L, Liguori G, James Copeland R, Del Villar Alvarez F, Jimenez A. High-intensity exercise to improve cardiorespiratory fitness in cancer patients and survivors: A systematic review and meta-analysis. Scand J Med Sci Sports. 2021 Feb;31(2):265-294. doi: 10.1111/sms.13861. Epub 2020 Nov 5. PMID 33098219
- [Result] Gouez M, Perol O, Perol M, Caux C, Menetrier-Caux C, Villard M, Walzer T, Delrieu L, Saintigny P, Marijnen P, Pialoux V, Fervers B. Effect of acute aerobic exercise before immunotherapy and chemotherapy infusion in patients with metastatic non-small-cell lung cancer: protocol for the ERICA feasibility trial. BMJ Open. 2022 Apr 7;12(4):e056819. doi: 10.1136/bmjopen-2021-056819. PMID 35393316